CLINICAL TRIAL: NCT07286916
Title: Impact of Guided Biofilm Therapy on Gingival Crevicular Fluid Epithelial and Mesenchymal Biomarkers in Periodontitis Patients: A Randomized Controlled Clinical Trial
Brief Title: Impact of Guided Biofilm Therapy on Epithelial and Mesenchymal Biomarkers in Periodontitis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Ibrahim Haider Sadeq, Dentist, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1108625
Record Dates: First submitted 2025-12-01; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Periodontitis
Keywords: Guided biofilm therapy; Gingival crevicular fluid; Epithelial Mesenchymal Transition; Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Intervention Model Description: The study is a 2 arm, split-mouth, double blinded, randomized clinical trial. The first group is control group will receive conventional NSPT (scaling & root surface debridement (RSD)), while the second group is the test group will be treated according to the GBT protocol.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional non-surgical periodontal therapy (NSPT) (Active Comparator): Control group
  Interventions: Procedure: Root surface debridement
- Guided Biofilm Therapy (GBT) (Experimental): Test group
  Interventions: Device: Guided Biofilm Therapy

INTERVENTIONS:
Procedure: Root surface debridement — Control group sites that will receive conventional NSPT will undergo supragingival debridement by using ultrasonic device at baseline. After one week, sites will receive root surface debridement (RSD) using area specific (Gracey) curettes (Medesy, Italy) according to the 24-hours protocol.
  Arms: Conventional non-surgical periodontal therapy (NSPT)
Device: Guided Biofilm Therapy — Test group sites will receive guided biofilm therapy (GBT) protocol using the Airflow Prophylaxis Master device by EMS which includes EMS DISCLOSING AGENT making the biofilm visible, EMS AIRFLOW combined with PLUS erythritol powder for removing biofilm, discoloration, and early calculus, PERIOFLOW removing the biofilm in deep periodontal pockets gently and thoroughly, and finally PIEZON PS for removing the remaining calculus.
  Arms: Guided Biofilm Therapy (GBT)

SUMMARY:
The goal of this clinical trial is to investigate the clinical and biochemical effects of the guided biofilm therapy protocol as an alternative to the conventional non-surgical periodontal therapy in patients with periodontitis. The main question it aims to answer is:

Does the guided biofilm therapy (GBT) protocol have an impact on gingival crevicular fluid (GCF) epithelial and mesenchymal biomarkers in patients with periodontitis?

All patients will be instructed to brush their teeth twice daily and will be supplied with the same type of toothpaste and toothbrush, with suitable interdental aids. All patients will be instructed to attend again after 7 days.

At baseline, full-mouth periodontal charting and radiographs will be obtained and after 1-hour, GCF samples will be collected from both test and control groups. Sites allocated to control group will undergo supragingival debridement by using ultrasonic device. After one week, the control group will receive RSD using area specific (Gracey) curettes (Medesy, Italy) according to the 24-hours protocol and will receive teeth polishing by using rubber polishing cups and tooth polishing paste, while the test group will receive a full GBT protocol which includes eight steps: (1) ASSESS, (2) DISCLOSE, (3) MOTIVATE, (4) AIRFLOW, (5) PERIOFLOW, (6) PIEZON PS*, (7) CHECK, and (8) RECALL. After finishing the treatment session, the patients will be asked to attend for follow up, clinical evaluation of PI, BOP, PPD, and CAL, and GCF samples collection after 1 month and 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects (>18 years).
2. Subjects are not currently under active periodontal therapy or joining other trial in the last 3 months.
3. Patients must be diagnosed with generalized unstable periodontitis with bilateral, symmetrical distribution of PPD ≥ 4mm and positive BOP.

   -

Exclusion Criteria:

1. Patients not diagnosed with periodontitis.
2. Patients consuming antibiotics.
3. Regular users of nonsteroidal anti-inflammatory drugs (NSAIDs).
4. Patients receiving periodontal treatment 3-months prior to the study.
5. Pregnant or mothers in a breastfeeding period.
6. Third molars and teeth with furcation involvement.
7. Patients taking antioxidant supplements.
8. Patients with heavy calculus that would prevent PerioPaper strips entrance to the periodontal pocket.
9. Patient with pulmonary diseases and with a history of allergy to erythritol.
10. Patients not willing to participate. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in probing pocket depth (PPD) | 3 months
  After treatment completion PPD ≤4mm with no BOP at 4mm pockets

SECONDARY OUTCOMES:
Clinical attachment level (CAL) | 3 months
Bleeding on probing (BOP) | 3 months
Plaque index (PI) | 3 months
Levels of gingival crevicular fluid (GCF) biomarkers | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- College of Dentistry, University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided